CLINICAL TRIAL: NCT05867225
Title: Onlay Synthetic Bioabsorbable Mesh Herniorrhaphy Versus Herniorrhaphy Only in the Primary Treatment of Large Hiatal Hernia: a Multicenter, Randomized, Parallel-group, Evaluator Blinded, Phase III Clinical Trial
Brief Title: Onlay Synthetic Bioabsorbable Mesh Herniorrhaphy Versus Herniorrhaphy Only in the Primary Treatment of Large Hiatal Hernia
Acronym: HIATUS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CHUBX 2021/23
Record Dates: First submitted 2022-12-30; First posted 2023-05-19 (Actual); Last update posted 2024-01-18 (Actual); Status verified 2024-01

CONDITIONS: Large Hiatal Hernia
Keywords: Large Hiatal Hernia; Recurrence; Surgery; Biosynthetic absorbable mesh
MeSH Terms: conditions — Recurrence

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Biosynthetic absorbable mesh (Experimental): Patients who have undergone hiatal surgery with use of a biosynthetic absorbable mesh
  Interventions: Procedure: Laparoscopic hiatal hernia repair
- No biosynthetic absorbable mesh (Sham Comparator): Patients who have undergone hiatal surgery without use of a biosynthetic absorbable mesh
  Interventions: Procedure: Laparoscopic hiatal hernia repair

INTERVENTIONS:
Procedure: Laparoscopic hiatal hernia repair — laparoscopic hiatal hernia repair has replaced the traditional laparotomic or thoracotomic approach, and has resulted in a reduction of length of hospital stay and morbidity, and increased patients' acceptance

SUMMARY:
The large hiatal hernia (LHH) now represents approximately 50% of laparoscopic antireflux surgical practice.

In a non-comparative retrospective study of 399 patients operated for LHH with onlay patch of a bioprosthetic absorbable (Gore® Bio-A® HH0710) mesh with a mean follow-up of 44 months, 16% had a symptomatic recurrence with 7,9% requiring reoperation, one patient had oesophageal stenosis. No comparative effectiveness data exist to date.

Hypothesis: the incidence of postoperative hiatus hernia would be reduced by the addition of biosynthetic absorbable mesh reinforcement to a standardized suture repair technique, as compared to laparoscopic repair without mesh, without increasing the risk of complications.

The main objective is to compare the radiologic recurrence rate at 2 years between standardized herniorrhaphy with onlay biosynthetic absorbable mesh repair versus standardized herniorrhaphy with no mesh in symptomatic LHH.

DETAILED DESCRIPTION:
The large hiatal hernia (LHH) now represents approximately 50% of laparoscopic antireflux surgical practice. Aging of the population and improvement of perioperative management may suggest that the number of these interventions will increase in the next few years. However, recurrence is common and has been described in up to 30% of patients who have undergone laparoscopic repair after a median follow up of 24 months.

The use of mesh reinforcement has been suggested to help preventing recurrence after LHH repair with non-absorbable and absorbable mesh.

In a non-comparative retrospective study of 399 patients operated for LHH with onlay patch of a bioprosthetic absorbable (Gore® Bio-A® HH0710) mesh with a mean follow-up of 44 months, 16% had a symptomatic recurrence with 7,9% requiring reoperation, one patient had oesophageal stenosis. No comparative effectiveness data exist to date.

Hypothesis: the incidence of postoperative hiatus hernia would be reduced by the addition of biosynthetic absorbable mesh reinforcement to a standardized suture repair technique, as compared to laparoscopic repair without mesh, without increasing the risk of complications.

The main objective is to compare the radiologic recurrence rate at 2 years between standardized herniorrhaphy with onlay biosynthetic absorbable mesh repair versus standardized herniorrhaphy with no mesh in symptomatic LHH.

The secondary objectives are :

* To compare the improvement of specific symptoms between two arms;
* To compare the Quality of life;
* To compare the complication rate and thecomplication severity according to the Clavien-Dindo classification;
* To assess the cost-effectiveness of standardized herniorrhaphy with onlay biosynthetic absorbable mesh repair as compared to standardized herniorrhaphy with no mesh, in symptomatic LHH, at 2 years, from the French Healthcare system point of view.

The expected benefits are :

* for the patient the diminution of LHH recurrence rate, quality of life improvement
* for Public health:
* Reducing the rate of reoperation for LHH;
* Reduction of healthcare costs due to a decrease in proton pump consumption and surgical re-interventions;
* The use of a synthetic bioprosthesis in laparoscopic surgery could be largely recommended and reimbursed either through the tariff related to the hospital stay (DRG tariff) or in additionto this tariff;
* Long term follow-up up to 5 years, could be obtained thanks to the use of French health insurance databases.

ELIGIBILITY:
Inclusion Criteria:

* Patient undergoing laparoscopic primary repair for symptomatic LHH. LHH is defined as a hiatal hernia larger than 5 cm in axial length as diagnosed at barium series and/or CT-scan with contrast swallow and/or CT-scan with contrast injection with axial reconstruction.
* Symptomatic hiatal hernia: heartburn and/or regurgitation and/or epigastric pain and/or dysphagia and/or anemia (if exclusion of other origin);
* Patient aged ≥ 18 years;
* Patient affiliated to a social security system or beneficiary of the same;
* Free written informed consent signed by the participant and the investigator (no later than the inclusion day and before performing any examination required for the study).

Exclusion Criteria:

* Patient undergoing reoperation for recurrent LHH repair;
* Emergency presentation needing an operation in a delay <6 hours;
* Asymptomatic hiatal hernia;
* American anesthesiologist score >3;
* Recurrent hiatal hernia and previous surgical interventions involving gastroesophageal junction;
* Brachyesophagus defined as the impossibility to achieve an intraabdominal length of the esophagus of at least 3cm after reduction of hernia contents and complete dissection and resection of the hernia sac;
* Previous major upper gastrointestinal surgery;
* Inability to perform primary closure of the crura;
* Pregnant or breast-feeding woman;
* Persons deprived of liberty or under guardianship or incapable of giving consent;
* Any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol or follow-up schedule, as assessed by investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 256 (Estimated)
Dates: Start 2024-01-15 (Actual); Primary Completion 2028-01-18 (Estimated); Study Completion 2028-01-18 (Estimated)

PRIMARY OUTCOMES:
Number of Large Hiatal Hernia recurrence | Month 24
  Radiologic recurrence will be identified at 24 months by an experienced radiologist blinded to the result of randomization and defined as the presence of any abdominal content located above the level of the diaphragm on CT-scan.

SECONDARY OUTCOMES:
Evaluation of Quality of life (QoL) by GIQLI, | Day 0
  GIQLI questionnaire includes 36 items relating to symptoms, physical status, emotions, social problems, and the effect of medical treatments. The score is between 0 and 144. The higher is the score, better is the quality of life.
Evaluation of Quality of life (QoL) by GIQLI, | Month 1
  GIQLI questionnaire includes 36 items relating to symptoms, physical status, emotions, social problems, and the effect of medical treatments. The score is between 0 and 144. The higher is the score, better is the quality of life.
Evaluation of Quality of life (QoL) by GIQLI, | Month 6
  GIQLI questionnaire includes 36 items relating to symptoms, physical status, emotions, social problems, and the effect of medical treatments. The score is between 0 and 144. The higher is the score, better is the quality of life.
Evaluation of Quality of life (QoL) by GIQLI, | Month 12
  GIQLI questionnaire includes 36 items relating to symptoms, physical status, emotions, social problems, and the effect of medical treatments. The score is between 0 and 144. The higher is the score, better is the quality of life.
Evaluation of Quality of life (QoL) by GIQLI, | Month 24
  GIQLI questionnaire includes 36 items relating to symptoms, physical status, emotions, social problems, and the effect of medical treatments. The score is between 0 and 144. The higher is the score, better is the quality of life.
Evaluation of Quality of life (QoL) by SF36 questionnaire | Day 0
  SF36 questionnaire consists of 36 items, including eight health-related scales: general physical condition, physical health role limitations, body pain, general health perception, vitality, social functioning, health role limitations psychic. The score is between 36 and 180. The higher is the score, better is the quality of life.
Evaluation of Quality of life (QoL) by SF36 questionnaire | Month 1
  SF36 questionnaire consists of 36 items, including eight health-related scales: general physical condition, physical health role limitations, body pain, general health perception, vitality, social functioning, health role limitations psychic. The score is between 36 and 180. The higher is the score, better is the quality of life.
Evaluation of Quality of life (QoL) by SF36 questionnaire | Month 6
  SF36 questionnaire consists of 36 items, including eight health-related scales: general physical condition, physical health role limitations, body pain, general health perception, vitality, social functioning, health role limitations psychic. The score is between 36 and 180. The higher is the score, better is the quality of life.
Evaluation of Quality of life (QoL) by SF36 questionnaire | Month 12
  SF36 questionnaire consists of 36 items, including eight health-related scales: general physical condition, physical health role limitations, body pain, general health perception, vitality, social functioning, health role limitations psychic. The score is between 36 and 180. The higher is the score, better is the quality of life.
Evaluation of Quality of life (QoL) by SF36 questionnaire | Month 24
  SF36 questionnaire consists of 36 items, including eight health-related scales: general physical condition, physical health role limitations, body pain, general health perception, vitality, social functioning, health role limitations psychic. The score is between 36 and 180. The higher is the score, better is the quality of life.
Evaluation of Quality of life (QoL) by EQ-5D-5L | Day 0
  EQ-5D-5L questionnaire comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems. The score is between 5 and 25. The lower is the score, better is the quality of life.
Evaluation of Quality of life (QoL) by EQ-5D-5L | Month 1
  EQ-5D-5L questionnaire comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems. The score is between 5 and 25. The lower is the score, better is the quality of life.
Evaluation of Quality of life (QoL) by EQ-5D-5L | Month 6
  EQ-5D-5L questionnaire comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems. The score is between 5 and 25. The lower is the score, better is the quality of life.
Evaluation of Quality of life (QoL) by EQ-5D-5L | Month 12
  EQ-5D-5L questionnaire comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems. The score is between 5 and 25. The lower is the score, better is the quality of life.
Evaluation of Quality of life (QoL) by EQ-5D-5L | Month 24
  EQ-5D-5L questionnaire comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems. The score is between 5 and 25. The lower is the score, better is the quality of life.
Evaluation of Quality of life (QoL) by EQ-VAS | Day 0
  EQ-VAS questionnaire asks patients to indicate their overall health on a vertical visual analogue scale, ranging from "worst possible" (score 0) to "best possible" health (score 100).
Evaluation of Quality of life (QoL) by EQ-VAS | Month 1
  EQ-VAS questionnaire asks patients to indicate their overall health on a vertical visual analogue scale, ranging from "worst possible" (score 0) to "best possible" health (score 100).
Evaluation of Quality of life (QoL) by EQ-VAS | Month 6
  EQ-VAS questionnaire asks patients to indicate their overall health on a vertical visual analogue scale, ranging from "worst possible" (score 0) to "best possible" health (score 100).
Evaluation of Quality of life (QoL) by EQ-VAS | Month 12
  EQ-VAS questionnaire asks patients to indicate their overall health on a vertical visual analogue scale, ranging from "worst possible" (score 0) to "best possible" health (score 100).
Evaluation of Quality of life (QoL) by EQ-VAS | Month 24
  EQ-VAS questionnaire asks patients to indicate their overall health on a vertical visual analogue scale, ranging from "worst possible" (score 0) to "best possible" health (score 100).
measurement of fever | Month 1
  measuring fever with a thermometer.Temperature is measured in degree Celsius (°C), between 34,7 and 40 °C.
measurement of fever | Month 6
  measuring fever with a thermometer.Temperature is measured in degree Celsius (°C), between 34,7 and 40 °C.
measurement of fever | Month 12
  measuring fever with a thermometer.Temperature is measured in degree Celsius (°C), between 34,7 and 40 °C.
measuring fever with a thermometer.Temperature is measured in degree Celsius (°C), between 34,7 and 40 °C. | Month 24
  measuring fever with a thermometer
measurement of weight | Day 0
  Measuring weight loss with a scale.The unit is kilogram. Weight change is between 30 and 150
measurement of weight | Month 1
  Measuring weight loss with a scale.The unit is kilogram. Weight change is between 30 and 150
measurement of weight | Month 6
  Measuring weight loss with a scale.The unit is kilogram. Weight change is between 30 and 150
measurement of weight | Month 12
  Measuring weight loss with a scale.The unit is kilogram. Weight change is between 30 and 150
measurement of weight | Month 24
  Measuring weight loss with a scale.The unit is kilogram. Weight change is between 30 and 150
measurement of blood pressure | Day 0
  Systolic and diastolic blood pressure are measured in millimeter of mercury (mm Hg). Systolic blood pressure is between 70 and 220 mm Hg. Diastolic blood pressure is between 20 and 160 mm Hg.
measurement of blood pressure | Month 1
  Systolic and diastolic blood pressure are measured in millimeter of mercury (mm Hg). Systolic blood pressure is between 70 and 220 mm Hg. Diastolic blood pressure is between 20 and 160 mm Hg.
measurement of blood pressure | Month 6
  Systolic and diastolic blood pressure are measured in millimeter of mercury (mm Hg). Systolic blood pressure is between 70 and 220 mm Hg. Diastolic blood pressure is between 20 and 160 mm Hg.
measurement of blood pressure | Month 12
  Systolic and diastolic blood pressure are measured in millimeter of mercury (mm Hg). Systolic blood pressure is between 70 and 220 mm Hg. Diastolic blood pressure is between 20 and 160 mm Hg.
measurement of blood pressure | Month 24
  Systolic and diastolic blood pressure are measured in millimeter of mercury (mm Hg). Systolic blood pressure is between 70 and 220 mm Hg. Diastolic blood pressure is between 20 and 160 mm Hg.

CONTACTS AND LOCATIONS:
Overall Officials: Caroline Gronnier, MD, PhD, Principal Investigator — University Hospital, Bordeaux
Locations (26):
- France (26):
  - CH de la Côte Basque, Bayonne
  - Hôpital Jean Minjoz, CHRU de Besançon, Besançon
  - Hôpital Cavale blanche, CHRU de Brest, Brest
  - Hôpital Côte de nacre, CHU Caen Normandie, Caen
  - Hôpital Estang, Clermont-Ferrand
  - Hôpital Louis-Mourier, AP-HP, Colombes
  - Hôpital Nord, CHU de Grenoble, La Tronche
  - Hôpital Claude Huriez, CHRU de Lille, Lille
  - Polyclinique du bois, Hôpital privé Le Bois, Lille
  - Hôpital Dupuytren 1, CHU de Limoges, Limoges
  - Hôpital de la Croix-Rousse, HCL, Lyon
  - Hôpital Saint Eloi, CHU de Montpellier, Montpellier
  - Hôpital Hôtel Dieu, CHU de Nantes, Nantes
  - Hôpital Archet, CHU de Nice, Nice
  - Hôpital Saint-Louis, AP-HP, Paris
  - Hôpital Saint-Antoine, AP-HP, Paris
  - DMU SAPERE, CHU Pitié-Salpêtrière APHP, Paris
  - Institut Mutualiste Montsouris, Paris
  - Hôpital Bichat, AP-HP, Paris
  - Hôpital du Haut Lévêque, Pessac
  - Hôpital Jean-Bernard, CHU de Poitiers, Poitiers
  - CH René-Dubos, Pontoise
  - CHU de Rennes, Site PONTCHAILLOU, Rennes
  - Hôpital Charles Nicolle, CHU de Rouen, Rouen
  - Hôpital Felix-Guyon, CHU de la Réunion, Saint-Paul
  - Hôpital Rangueil, CHU de Toulouse, Toulouse

IPD SHARING:
Plan to Share IPD: No